CLINICAL TRIAL: NCT07328906
Title: Steroid Treatment to Prevent Thoracic Endovascular Aortic Repair Postimplantation Syndrome (STOP TEVAR PIS): A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Steroid Treatment to Prevent Thoracic Endovascular Aortic Repair Postimplantation Syndrome
Acronym: STOP TEVAR PIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Igor Koncar, Vascular surgeon, MD, Ph.D., University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STOP TEVAR PIS
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postimplantation Syndrome; Myocardial Injury; MACE; Mortality
Keywords: postimplantation syndrome; methylprednisolone; TEVAR; myocardial injury; MACE; mortality
MeSH Terms: interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MP (experimental group) (Experimental): Intervention: methylprednisolone preoperatively 30 mg/kg.
  Patients in the MP group will receive 30 mg/kg of methylprednisolone, dissolved in 100 mL of saline, via a 30-minute slow intravenous infusion.
  Interventions: Drug: Methylprednisolone (MP)
- Control group (placebo) (Placebo Comparator): Patients randomized to the placebo group will receive 100 mL of physiological solution two hours prior to the intervention.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Drug: Methylprednisolone (MP) — Patients in the MP group would receive 30 mg/kg of methylprednisolone, dissolved in 100 mL of saline, via a 30-minute slow intravenous infusion.
  Arms: MP (experimental group)
Drug: Placebo (saline) — Patients randomized to the placebo group would receive 100 mL of physiological solution two hours prior to the intervention.
  Arms: Control group (placebo)

SUMMARY:
Postimplantation syndrome (PIS) is a common and clinically important complication following thoracic endovascular aortic repair (TEVAR). PIS is characterized by a strong systemic inflammatory response to the stent-graft implantation and is manifested by flu-like symptoms, which include fever, increased white blood count, increased levels of acute phase proteins, and fatigue, but without a clear inflammatory and infective cause. Besides, it has been demonstrated that PIS is associated with prolonged hospital stay and increased risk for postoperative complications, including acute kidney injury, postoperative delirium, and increased postoperative pain scores. Recently, there has been increasing evidence that PIS is associated with an increased risk of major adverse cardiac events (MACE) and perioperative myocardial injury. Observational studies suggest that preoperative administration of glucocorticoids may decrease the incidence of PIS after TEVAR and EVAR procedures. However, to date, there are no randomised trials that have investigated whether preoperative administration of glucocorticoids can reduce the incidence of PIS and its associated poorer treatment outcomes following TEVAR. This randomized controlled trial was designed to investigate the effect of glucocorticoid administration on reducing the incidence and improving the outcome of patients who develop PIS after TEVAR.

DETAILED DESCRIPTION:
Postimplantation syndrome (PIS) is a common and clinically important complication following thoracic endovascular aortic repair (TEVAR). Although PIS incidence following endovascular procedures varies widely from 2% to 100%, (1, 2) according to the majority of studies investigating this topic, this entity may be noted in approximately one-third of patients following TEVAR. (3-5) PIS is characterized by a strong systemic inflammatory response to the stent-graft implantation and is manifested by flu-like symptoms, which include fever, increased white blood count, increased levels of acute phase proteins, and fatigue, but without a clear inflammatory and infective cause. Besides, it has been demonstrated that PIS is associated with prolonged hospital stay and increased risk for postoperative complications, including acute kidney injury, postoperative delirium, and increased postoperative pain scores. Recently, there has been increasing evidence that PIS is associated with an increased risk of major adverse cardiac events (MACE) and perioperative myocardial injury, which may have significant long-term consequences. (6, 7) Despite all this, the pathohistological mechanisms of PIS have not been fully elucidated, and available therapeutic options for prevention and treatment are limited. (8) It has been demonstrated that the administration of glucocorticoids can contribute to reducing the incidence of PIS after endovascular procedures on the abdominal aorta (EVAR), due to their potent anti-inflammatory effects that modulate the body's response to stent-graft implantation. (9, 10) Since PIS is a form of non-specific systemic inflammatory reaction to a foreign body, accompanied by mechanical damage to the endothelium, glucocorticoids can act preventively by inhibiting the production of cytokines (e.g., IL-6, TNF-α), reducing capillary permeability, stabilizing the leukocyte membrane, and reducing the expression of adhesion molecules. Observational studies suggest that preoperative administration of methylprednisolone or hydrocortisone may lead to a reduction in the incidence of PIS, lower CRP levels, and a shorter duration of febrile response after TEVAR and EVAR procedures. (11, 12) However, for patients undergoing TEVAR, contemporary literature data are limited and originate from observational studies. To date, there are no high-quality clinical studies that have investigated whether preoperative administration of glucocorticoids can reduce the incidence of PIS and its associated poorer treatment outcomes following TEVAR. This randomized controlled trial was designed to investigate the effect of glucocorticoid administration on reducing the incidence and improving the outcome of patients who develop PIS after TEVAR.

The aims of the study are: 1. to examine whether preoperative administration of methylprednisolone (in a single bolus dose of 30 mg/kg of body weight) reduces the frequency of post-implantation syndrome in the first 5 days after TEVAR; 2. to examine the impact of preoperative administration of methylprednisolone on reducing the incidence of myocardial injury immediately postoperatively, after TEVAR; 3. to assess the frequency of MACE during hospitalization, one month, and two years after the TEVAR procedure; 4. to assess the degree of aortic remodeling by CT after one month and two years after TEVAR; 5. evaluate the frequency of other surgical and non-surgical complications, the intensity of postoperative pain (measured using the Numeric Rating Scale - NRS, during 48 hours postoperatively), as well as the length of stay in the Intensive Care Unit and the length of hospital stay; 6. to estimate 30-day and total 2-year mortality.

This double-blind, randomized, placebo-controlled study will be conducted at 3 international centers. The estimated duration of the study is 12 months, followed by a period of short-term (one month) and long-term (two years) follow-up. The study will include consecutive patients older than 18 years who undergo elective TEVAR procedures for aortic dissection type B or thoracoabdominal aortic aneurysm, in whom, according to current guidelines, an indication for endovascular treatment has been established, (13) who are capable of giving informed consent, and who are estimated to be available for long-term follow-up. Exclusion criteria would include emergency procedures, the existence of severe renal insufficiency (serum creatinine >176 µmol/L or estimated glomerular filtration rate < 30 mL/min/1.73 m2), severe liver insufficiency (ALT value more than twice the upper limit or bilirubin levels more than twice the reference values), uncontrolled diabetes mellitus (fasting glycemia above 13.9 mmol/L, i.e. the value glycosylated hemoglobin over 8.5%), existence of active infection or sepsis, autoimmune disease, chronic pain syndromes, proven allergy to methylprednisolone, existence of gastric or duodenal ulcer, immunosuppressive or chemotherapy in the previous three months, active malignant disease, genetic diseases of connective tissue, pregnancy, critical lower limb ischemia, previous endovascular procedure on the aorta, preoperative administration of corticosteroids for any reason, significantly impaired cognitive status or psychiatric illness, acute peri/myocarditis, advanced heart failure, as well as voluntary refusal to participate in the study. Body temperature would be measured three times per day during the first five postoperative days.

Randomization: Subjects will be randomized into two groups, in a 1:1 ratio, namely: 1) experimental (methylprednisolone, MP) group, and 2) control (placebo) group. Double-blind randomization would be performed using computer-generated randomization codes by an investigator, not directly participating in any form of the treatment of patients included in the study. The assignment of subjects to one of the groups would be revealed only on the day of the procedure, two hours before induction of anesthesia. At that time, patients in the MP group would receive 30 mg/kg of methylprednisolone, dissolved in 100 mL of saline, via slow intravenous infusion lasting 30 minutes. Patients randomized to the placebo group would receive 100 mL of physiological solution two hours prior to the intervention. Both groups would receive a selective proton pump inhibitor (pantoprazole 40 mg IV, twice daily), starting the day before surgery. All other aspects of perioperative treatment will be the same for subjects from both groups and standardized according to institutional protocols. Patients will be operated under general endotracheal anesthesia or under local infiltrative anesthesia with sedation, and surgical TEVAR protocols and anesthesia protocols will be uniformly standardized. Half an hour before the start of the TEVAR procedure, all patients would receive antibiotic prophylaxis (ceftriaxone 2g, bolus dose) and ondansetron (4 mg, to prevent postoperative nausea and vomiting). At the end of the procedure and during the first three postoperative days, patients would be monitored to assess neurological status (including the appearance of spinal cord ischemia) every 2-4 hours. In the event of symptoms/signs indicating spinal cord ischemia, a catheter for CSF drainage would be placed, and the CSF pressure would be maintained in the range of 10-12 mmHg, with a maximum drainage of 20 ml/h. Also, in patients with a high risk for the occurrence of spinal cord ischemia (overlapping of the thoracic aorta over 15-20 mm in length, previous open aortic surgery, compromised pelvic perfusion - stenosed or occluded common or internal iliac arteries, stenosed or occluded vertebral arteries, planned overlap of the left subclavian artery, or when the patient is assessed as high-risk by the operator) the catheter would be placed preoperatively (prophylactically). Peripheral venous blood would be sampled from all patients for the evaluation of biochemical parameters of interest, during first five postoperative days, which, in addition to the standard necessary analyses, would include: the total number of leukocytes, the level of C-reactive protein, fibrinogen, D-dimer, and high-sensitivity troponin I (hs-TnI) the day before TEVAR, and the first three days after the procedure (6h, 24h and 72h following TEVAR).

Data collection: Basic demographic, anthropometric, and clinical data of interest (including data on current illness, comorbidities, smoking status, preoperative chronic therapy, as well as standard laboratory and coagulation parameters) would be collected through patient interviews and/or review of medical records. Data related to the intraoperative and postoperative course (including the length of stay in the ICU, postoperative complications, intrahospital mortality, etc.) will be obtained based on medical documentation and the database included in the daily work of the Clinic. Data related to the period of short-term (one month) and long-term (one year after TEVAR) threat would be collected through interviews and medical documentation at regularly scheduled follow-up examinations. Post-implantation syndrome would be defined as the occurrence of elevated body temperature (>38.0°C), with the presence of leukocytosis (12,000/mm³), and an increase in the level of C-reactive protein (>10g/L) during the first three days postoperatively, despite negative blood cultures. (2) MACE events would be defined as a composite outcome that includes the occurrence of myocardial infarction, acute heart failure, malignant rhythm disorders, and cardiovascular death. Myocardial injury would imply an increase in the level of hs-TnI above the 99th percentile of the upper reference limit, i.e. in patients with chronic myocardial injury (initially elevated values of this cardiac biomarker), only acute myocardial injury will be considered - an increase and/or decrease of more than 20% from the basal value, without clinical signs of acute myocardial ischemia. (14) Data related to pain intensity would be collected at regular intervals (once during 24h), the first three postoperative days, whereby the patient would answer a question about pain intensity on a scale from 0 (no pain) to 10 (worst possible pain) according to the Numerical Pain Scale. Reintervention would be defined as reoperation of a given patient within the first 48 hours after the operation due to the occurrence of acute bleeding or thrombosis. Postoperative pulmonary complications would be defined as the occurrence of respiratory disorders in the immediate postoperative period, namely: hypoxemia, hypercapnia, acute bronchospasm, laryngospasm, pneumothorax, pulmonary edema, pneumonia, pleural effusion, prolonged mechanical lung ventilation (>48h), acute respiratory distress syndrome, and the need for re-intubation of the trachea due to respiratory insufficiency. Neurological complications would include cerebrovascular insult, transient ischemic attack, and other neurological disorders. Complications from the digestive system would include diarrhea, hematemesis, or melena. The diagnosis of postoperative acute renal failure would be made in accordance with the KDIGO guidelines (Kidney Disease: Improving Global Outcomes) as an increase in the level of serum creatinine by ≥ 26.5 μmol/L during 48h, or an increase in the initial value of creatinine by ≥ 1.5 times that is known or assumed to have occurred during the previous seven days, or diuresis < 0.5 ml/kg/h during six hours. (15) Local wound infection would be defined as the appearance of redness, pain, and/or drainage at the incision site, with an increase in the infection parameters, with or without a temperature > 38°C. Postoperative hemodynamic instability is defined as the occurrence of hypertension (an increase in systolic blood pressure above 180 mmHg, requiring therapeutic measures) and/or hypotension (a decrease in systolic blood pressure below 90 mmHg, also requiring therapeutic measures), with or without cardiac rhythm disturbances. For this study, the occurrence of postoperative delirium will be considered, as defined by the American Psychiatric Association (APA) DSM-5 criteria from 2013, and the existence of documentation on the use of neuroleptics. (16) The length of stay in the Intensive Care Unit would mean the time from leaving the operating room to the discharge of the patient to semi-intensive care, while the length of hospitalization would be defined as the time elapsed from admission to hospital discharge.

Sample size and power calculation: Sample size estimation was based on the expected incidence of PIS and the desired therapeutic effect of the intervention. According to the available literature, the incidence of PIS after TEVAR is approximately 30% in patients not receiving anti-inflammatory prophylaxis. The use of methylprednisolone is expected to lead to a 50% relative reduction in the incidence of PIS, resulting in a 15% absolute frequency in the experimental group. To observe the desired difference between the groups with a probability of 80%, at a significance level of 5%, and an equal distribution of patients in both groups (1:1), it was calculated that the required sample size is a total of 158 subjects (79 per group). Considering the possibility of withdrawal, loss during the follow-up period, or other reasons for exclusion, which could result in up to 10% of subjects being excluded from the study, the definitive sample size is 174 patients (87 per group).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted due to endovascular treatment of aortic dissection type B or thoracoabdominal aortic aneurysm in whom elective, open repair is planned.
* Patients capable of giving informed consent.
* Patients who are estimated to be available for long-term follow-up.

Exclusion Criteria:

* emergency procedures, the existence of severe renal insufficiency (serum creatinine >176 µmol/L or estimated glomerular filtration rate < 30 mL/min/1.73 m2), severe liver insufficiency (ALT value more than twice the upper limit or bilirubin levels more than twice the reference values), uncontrolled diabetes mellitus (fasting glycemia above 13.9 mmol/L, i.e. the value glycosylated hemoglobin over 8.5%), existence of active infection or sepsis, autoimmune disease, chronic pain syndromes, proven allergy to methylprednisolone, existence of gastric or duodenal ulcer, immunosuppressive or chemotherapy in the previous three months, active malignant disease, genetic diseases of connective tissue, pregnancy, critical lower limb ischemia, previous endovascular procedure on the aorta, preoperative administration of corticosteroids for any reason, significantly impaired cognitive status or psychiatric illness, acute peri/myocarditis, advanced heart failure, as well as voluntary refusal to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of PIS | 5 days postoperatively
  Post-implantation syndrome would be defined as the occurrence of elevated body temperature (>38.0°C), with the presence of leukocytosis (>12,000/mm³), and an increase in the level of C-reactive protein (>10g/L) during the first five days postoperatively, despite negative blood cultures.

SECONDARY OUTCOMES:
incidence of myocardial injury | first 3 days postoperatively
  Myocardial injury would be defined as an increase in the level of hs-TnI above the 99th percentile of the upper reference limitwithout clinical signs of acute myocardial ischemia, during the first three postoperative days.
incidence of MACE | 2 years postoperatively
  MACE events would be defined as a composite outcome that includes the occurrence of myocardial infarction, acute heart failure, malignant rhythm disorders, and cardiovascular death during two years after TEVAR.
intensity of postoperative pain | two days postoperatively
  The intensity of postoperative pain will be measured using the Numeric Rating Scale - NRS, during 48 hours postoperatively.
degree of aortic remodeling | one month and two years postoperatively
  Degree of aortic remodeling will be assessed based on CT evaluation of the aorta) one month and two years after TEVAR
30-day mortality rate | one month postoperatively
  30-day mortality would refer to any lethal outcome (due to any cause), that would occur 30 days following surgery.
long-term mortality rate | two years after TEVAR
  Long-term mortality would refer to any lethal outcome (due to any cause), that would occur 2 years following TEVAR.

OTHER OUTCOMES:
surgical complications | 30 days after TEVAR
  Postoperative surgical complications will be defined as complications related to the surgical procedure within 30 days after the operation.
non-surgical complications | 30-days after TEVAR
  Postoperative non-surgical complications will be defined as complications which are not related to surgical procedures/techniques and are related to patients' physiological status or comorbidities.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Vascular and Endovascular Surgery, University Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 16. American Psychiatric Association. American Psychiatric Association: Diagnostic and Statistical Manual of Mental Disorders. 2013;5th ed. Arlington, VA.
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; ESC Scientific Document Group. Fourth universal definition of myocardial infarction (2018). Eur Heart J. 2019 Jan 14;40(3):237-269. doi: 10.1093/eurheartj/ehy462. No abstract available. PMID 30165617
- [Background] Upchurch GR Jr, Escobar GA, Azizzadeh A, Beck AW, Conrad MF, Matsumura JS, Murad MH, Perry RJ, Singh MJ, Veeraswamy RK, Wang GJ. Society for Vascular Surgery clinical practice guidelines of thoracic endovascular aortic repair for descending thoracic aortic aneurysms. J Vasc Surg. 2021 Jan;73(1S):55S-83S. doi: 10.1016/j.jvs.2020.05.076. Epub 2020 Jul 3. PMID 32628988
- [Background] Zhu Y, Luo S, Ding H, Liu Y, Huang W, Xie N, Li J, Xue L, Luo J. Predictors associated with an increased prevalence of postimplantation syndrome after thoracic endovascular aortic repair for type B aortic dissectiondagger. Eur J Cardiothorac Surg. 2019 May 1;55(5):998-1005. doi: 10.1093/ejcts/ezy379. PMID 30521031
- [Background] 11. Dworak T, Mäurer L, Kolbenschlag J, Bockler D, Kotelis D. Preoperative corticosteroids in EVAR and TEVAR - is there an impact on postimplantation syndrome? Vascular. 2020;28(6):648-654.
- [Background] 10. Becquemin JP, Kelly P, Zubilewicz T, Desgranges P, Allaire E, Kobeiter H. Postimplantation syndrome after endovascular aneurysm repair: incidence, predictive factors, and outcome. Eur J Vasc Endovasc Surg. 2003;25(2):139-145.
- [Background] 9. Kobayashi K, Sato M, Inoue M, Shibata Y, Asai Y. Steroid pretreatment attenuates the systemic inflammatory response after endovascular aneurysm repair. J Vasc Surg. 2015;61(1):127-134.
- [Background] 8. Soares Ferreira R, Bastos Gonçalves F. Postimplantation syndrome after endovascular aneurysm repair. In: Koncar I, editor. Abdominal Aortic Aneurysm - From Basic Research to Clinical Practice. IntechOpen; 2018.
- [Background] Mannina C, Kini A, Carbone A, Neibart E, Bossone E, Prandi FR, Tadros R, Esposito G, Erbel R, Sharma SK, Lerakis S. Management of Systemic Inflammatory Response Syndrome After Cardiovascular Interventions. Diagnostic, Prognostic, and Therapeutic Implications. Am J Cardiol. 2024 Jun 15;221:84-93. doi: 10.1016/j.amjcard.2024.04.007. Epub 2024 Apr 20. PMID 38649128
- [Background] Sousa J, Vilares AT. Postimplantation Syndrome Is Not Associated with Myocardial Injury after Noncardiac Surgery after Endovascular Aneurysm Repair. Ann Vasc Surg. 2020 Oct;68:275-282. doi: 10.1016/j.avsg.2020.04.014. Epub 2020 Apr 25. PMID 32339692
- [Background] 5. Lee S, Kim H, Park J, Moon JY, Yang JH, Chung J, et al. Risk prediction and prognostic analysis of post-implantation syndrome after thoracic endovascular aortic repair. J Endovasc Ther. 2023;30(4):536-43.
- [Background] Wu Q, He J, Li H, Xie L, Zeng W, Lin X, Qiu Z, Chen L. Outcomes of post-implantation syndrome after endovascular repair for Stanford type B aortic dissection. J Vasc Surg. 2024 Jun;79(6):1326-1338. doi: 10.1016/j.jvs.2024.01.200. Epub 2024 Jan 28. PMID 38286152
- [Background] Wang B, Miao M, Shi Q, Xian H, Cao Y, Wang X. Impact of post-implantation syndrome on outcomes in acute type B aortic syndrome patients undergoing endovascular repair. Vasa. 2024 Jan;53(1):53-60. doi: 10.1024/0301-1526/a001102. Epub 2023 Nov 15. PMID 37965717
- [Background] de la Motte L, Kehlet H, Vogt K, Nielsen CH, Groenvall JB, Nielsen HB, Andersen A, Schroeder TV, Lonn L. Preoperative methylprednisolone enhances recovery after endovascular aortic repair: a randomized, double-blind, placebo-controlled clinical trial. Ann Surg. 2014 Sep;260(3):540-8; discussion 548-9. doi: 10.1097/SLA.0000000000000895. PMID 25115430
- [Background] Melissano G, Tshomba Y, Rinaldi E, Chiesa R. Initial clinical experience with a new low-profile thoracic endograft. J Vasc Surg. 2015 Aug;62(2):336-42. doi: 10.1016/j.jvs.2015.02.049. Epub 2015 Apr 30. PMID 25935267